CLINICAL TRIAL: NCT01127217
Title: The Multicenter, Randomized, Double Blind Phase 3 Clinical Trial to Compare Efficacy and Safety of Combination of Amlodipine and Losartan Compared to Amlodipine Monotherapy in Patients With Stage 2 Hypertension
Brief Title: Efficacy/Safety of Amlodipine Plus Losartan Versus Amlodipine in Patients With Stage 2 Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-ALOS-303
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Hypertension
Keywords: amlodipine; losartan; hypertension; stage 2
MeSH Terms: conditions — Hypertension | interventions — amlodipine-losartan drug combination; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- amlodipine/losartan (Experimental)
  Interventions: Drug: amlodipine/losartan
- amlodipine (Active Comparator)
  Interventions: Drug: amlodipine

INTERVENTIONS:
Drug: amlodipine/losartan — amlodipine 5mg/losartan 50mg, amlodipine 10mg/losartan 50mg (+HCTZ 12.5mg)
  Other Names: amosartan
  Arms: amlodipine/losartan
Drug: amlodipine — amlodipine 5mg, amlodipine 10mg (+ HCTZ 12.5mg)
  Other Names: amodipin(amlodipine camsylate)
  Arms: amlodipine

SUMMARY:
The purpose of this study is to evaluate the blood pressure lowering effects of an amlodipine/losartan combination treatment and amlodipine monotherapy for treatment of Stage 2 hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 aged or over
* Patients with blood pressure measured at Visit 1; MSSBP≤180mmHg and MSDBP≤110 mmHg if on anti-hypertensive drugs, 160mmHg≤MSSBP≤199mmHg and 80mmHg≤MSDBP≤119mmHg if not on anti-hypertensive drugs
* Patients with blood pressure measured at Visit 2 were 160mmHg≤MSSBP≤199mmHg and 80mmHg≤MSDBP≤119mmHg

Exclusion Criteria:

* Inability to stop all prior anti-hypertensive drugs safely during wash out period of 3 to 7 days
* ≥ sitSBP 20mmHg or ≥ sitDBP 10mmHg of variation in three measurements from the reference arm selected at Screening
* History of hypersensitivity to dihydropyridines, angiotensin II receptor blockers or thiazide diuretics
* Secondary hypertension or suspected to be
* Continuously took medicinal drugs that might affect blood pressure rather than anti-hypertensive drugs more than 3 months
* Type 2 diabetes mellitus which is not controlled or with type 1 diabetes mellitus
* History of severe neurovascular disease, severe heart disease
* Known as moderate or malignant retinopathy.
* Renal diseases; serum creatinine ≥ 2mg/dl
* Hepatic diseases; increase in ALT or AST ≥ 2xUNL
* Anuria
* Hyponatremia/hypokalemia or hypercalcemia
* Active Gout
* Surgical or medical diseases which might significantly change ADME of medicines
* History of malignant tumor
* Autoimmune diseases
* History of alcohol or drug abuse
* Positive to pregnancy test, nursing mother, woman with an intention of pregnancy
* Considered inappropriate to participate in the clinical trial with any reason, based on investigator's decision

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in MSSBP | Baseline, Week 6

SECONDARY OUTCOMES:
Change from baseline in MSSBP | Baseline, Week 2 and 8
Change from baseline MSDBP | Baseline, Week 2, 6, and 8
Blood pressure responder rate | Baseline, Week 2, 6, 8
  Rate of patients who achieved target blood pressure (MSSBP < 140 mmHg or MSDBP < 90 mmHg), or MSSBP decrease > 20 mmHg from baseline or MSDBP decrease > 10 mmHg from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- 8 Sites, Seoul, South Korea

REFERENCES:
- [Derived] Kim SH, Ryu KH, Lee NH, Kang JH, Kim WS, Park SW, Lee HY, Kim JJ, Ahn YK, Suh SY. Efficacy of fixed-dose amlodipine and losartan combination compared with amlodipine monotherapy in stage 2 hypertension: a randomized, double blind, multicenter study. BMC Res Notes. 2011 Oct 28;4:461. doi: 10.1186/1756-0500-4-461. PMID 22035131